CLINICAL TRIAL: NCT07052240
Title: GTK-UNI: Effectiveness of a Suicide Prevention Gatekeeper Program in the University Setting
Brief Title: Implementation of a Suicide Prevention Gatekeeper Program in the University Setting
Acronym: GTK-UNI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, María Sandra Pérez Rodríguez, Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-PSILOG-3746002
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Suicide Prevention; Suicide Awareness; Suicide Behavior
Keywords: Suicide Prevention; Gatekeeper Training; University Students; Mental Health Literacy; Suicide Awareness; Stigma Reduction; Help-Seeking Behavior
MeSH Terms: conditions — Suicide Prevention; Help-Seeking Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial, efficacy Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gatekeeper Immediate Training Group (GTK-IG) (Experimental): Participants in this arm are university students who will receive the Gatekeeper Immediate Training (GTK-IG) during the main phase of the study, either face-to-face or online. The training includes two 3-hour sessions held one week apart, covering six structured modules: (1) Introduction to suicidal behavior (key concepts, myths, and statistics); (2) Warning signs and risk/protective factors based on the interpersonal theory of suicide; (3) Suicide crisis intervention and first aid techniques; (4) Safety planning and identification of local support resources; (5) Ethical considerations and self-care for gatekeepers; and (6) Practical skill application through simulations and discussion. Participants will complete pre- and post-intervention evaluations (T0, T1), as well as a follow-up assessment two-three months after T1 (T2), and 9-12 months after T1, followed by a booster session and a focus group to explore skill retention and real-world application.
  Interventions: Behavioral: Gatekeeper Training Program (GTK)
- Delayed Gatekeeper Training (GTK-DG) (No Intervention): Participants in this arm will not receive any intervention during the main phase of the study. They will follow the same assessment schedule as the intervention group at three time points: before the program (T0), immediately after the intervention group completes training (T1), and two months later (T2). After completing the T2 evaluation, participants in this group will be offered the Delayeed Gatekeeper Training (GTK-DG) under the same conditions as the intervention group (face-to-face or online). This waitlist design ensures ethical access to the program while allowing for comparisons between trained and untrained participants during the primary analysis period.

INTERVENTIONS:
Behavioral: Gatekeeper Training Program (GTK) — Behavioral: Gatekeeper Training Program (GTK-UNI)
  The GTK program is a suicide prevention intervention for university students. It includes two sessions of 3 hours each (total: 6 hours), delivered over one week, either face-to-face or online. Content is organized into six modules:
  1. Introduction to suicidal behavior.
  2. Warning signs and risk/protective factors.
  3. Crisis intervention and suicide first aid.
  4. Safety planning and community resources.
  5. Ethics and gatekeeper self-care.
  6. Practical simulations and skill application.
  The program includes interactive exercises, role-plays, take-home materials, and a booster session plus a focus group at the 2-month follow-up.
  Arms: Gatekeeper Immediate Training Group (GTK-IG)

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of a suicide prevention training program (Gatekeepers) tailored to university students in Spain. The main questions it aims to answer are:

* Does the training program improve suicide-related knowledge, attitudes, perceived behavioral control, and gatekeeper behaviors among students?
* Are there differences in training outcomes by gender, and how do they affect program engagement and effectiveness? Researchers will compare a Immediate Intervention Group (GTK-IG), which will receive the full training immediately, with a 2) the Delayed Intervention Group (GTK-DG), which will be a waitlist control during the first phase of the study, to evaluate the program's short- and medium-term impact, using both in-person and online formats. which will be a waitlist control during the first phase of the study.

Participants will:

* Be randomly assigned to the intervention or control group, choosing between in-person or online training
* Complete online surveys at three timepoints: before the program (T0), immediately after (T1), 2-3 months later (T2), and 9-12 months follow-up (T3).
* Attend two 3-hour training sessions covering key suicide prevention competencies
* Participate in a follow-up session with focus group discussion to qualitatively assess retention and use of learned skills
* Complete validated questionnaires on suicide prevention literacy, attitudes, stigma, and self-reported gatekeeper behaviors This trial includes validation of the Spanish versions of the WISE (Willingness to Intervene Against Suicide Enhanced Questionnaire) and ACT as Gatekeeper measures. The study is registered at ClinicalTrials.gov and follows CONSORT and SPIRIT guidelines. Ethical approval was granted by the Human Research Ethics Committee at the University of Valencia.

DETAILED DESCRIPTION:
Title: Effectiveness of a Multicenter Suicide Prevention Gatekeeper Program for Students at Spanish Universities (GTK-UNI)

Background and Rationale:

Suicide is a leading cause of death among young adults worldwide, and university students represent a particularly vulnerable population due to psychosocial, academic, and transitional stressors. Despite the growing recognition of the importance of suicide prevention, few evidence-based interventions have been adapted for university environments in Spain. Gatekeeper Training (GKT) programs are short interventions designed to equip non-specialists with the ability to recognize warning signs, intervene appropriately, and refer at-risk individuals to professional support. This project, titled GTK-UNI, aims to develop, implement, and rigorously evaluate the effectiveness of a Gatekeeper Training program adapted to Spanish university settings.

Study Objectives:

The main objective of this multicenter randomized controlled trial (RCT) is to evaluate the effectiveness of a suicide prevention Gatekeeper program delivered to university students. The program will be tested both in online and face-to-face formats to determine its utility, scalability, and long-term impact. Specific aims include:

Designing a structured and culturally relevant GKT program for university students in Spain.

Validating two measurement tools in Spanish: the Willingness to Intervene Against Suicide Enhanced Questionnaire (WISE) and the ACT as Gatekeeper questionnaire.

Implementing the program in both in-person and online formats to ensure accessibility.

Measuring the impact of the training on knowledge, attitudes, perceived control, and actual gatekeeper behaviors, with gender-stratified analyses.

Evaluating participants' adherence to and satisfaction with the program, identifying gender-related barriers and facilitators to participation.

Collecting qualitative data through focus groups to explore how gender norms influence program engagement and effectiveness.

Disseminating results to support gender-sensitive suicide prevention strategies in educational and mental health policy.

Contributing to translational research by developing a validated guide for university-level suicide prevention planning.

Methods:

This is a multicenter, two-arm, randomized controlled trial with a waitlist control group. Participants are university students (age ≥18) from multiple Spanish universities, recruited via university mailing lists, social media, student associations, and institutional partnerships. Recruitment materials clarify that the training is a suicide prevention initiative and outline the voluntary nature of participation.

Randomization and Conditions:

After providing informed consent, participants are randomly assigned to one of two groups:

Intervention group (GTK-IG): Receives the Gatekeeper Training immediately, either in online or face-to-face format, depending on their preference.

Delayed Intervention Group (GTK-DG): which will be a waitlist control during the first phase of the study and will receive the interventions after T2 (2-3 months later).

Training Format and Content:

The GTK-UNI program consists of 6 modules delivered in two 3-hour sessions over two weeks. Modules include:

Introduction to suicidal behavior and epidemiology

Recognition of warning signs and risk/protective factors

Crisis intervention and suicide first aid strategies

Safety planning and community resources

Ethics and self-care for gatekeepers

Practical evaluation and case simulation

Evaluation Timeline:

T0 (Baseline): Online survey before intervention

T1 (Post-intervention): Immediately after last session (two weeks after T0)

T2 (Follow-up): To be conducted 2 months after T1, with a booster session and focus group for GTK-GE participants scheduled approximately 2.5 months after T0.

T3 (Follow up 2): 9-12-month after T1.

After each session: Assessments will be also administered to monitor progressive skill acquisition.

Control group receives the training after T2 (approximately 2.5-3 months after T0)

Instruments:

Primary outcome measures include:

WISE Questionnaire (Aldrich & Cerel, 2024): Measures attitudes, norms, perceived control, and intention to intervene.

ACT as Gatekeeper (Nozawa et al., 2020): Evaluates actual gatekeeper behaviors.

Secondary outcomes:

LOSS-SF (Calear et al., 2022): Assesses suicide literacy. SOSS-SF (Batterham et al., 2012): Measures stigma toward suicide. PHQ-9 (Kroenke et al., 2001): Assesses depressive symptoms. Additional variables include emotional burden, satisfaction, gender, and open-ended responses on program perception.

Rosenbertg self steem (Rosenberg, 1965) Program satisfaction and perceived utility. Ad hoc questions. Suicidal behavior (self and others). Ad hoc questions. Intersession skill monitoring: ad hoc questions.

Ethical Considerations:

The study protocol was approved by the Human Research Ethics Committee of the University of Valencia (ID: UV-INV_ETICA-3746002). The project adheres to the Declaration of Helsinki, the Madrid Declaration of the World Psychiatric Association, and national ethical standards. All participants will provide informed consent and retain the right to withdraw at any time. Data will be anonymized and securely stored, with no sharing of personal information with third parties.

If participants report emotional distress or indicate prior suicidal behavior as a motivation for joining, LIme Survey platform triggers an emergency screen with contact information for psychological services and crisis helplines. Professional referral may be offered as needed.

Sample Size and Power Calculation:

Sample size calculations were based on previous studies evaluating GTK, assuming medium effect sizes for attitudinal and self-efficacy outcomes (Cohen's d = 0.50), a power of 0.80, and α = 0.05. Allowing for an estimated attrition rate of 20-25%, the target sample size was set to ensure sufficient statistical power for mixed-model and between-group analyses. The final recruitment goal was approximately 420 participants, distributed evenly between experimental conditions.

Data Collection and Analysis:

All assessments are administered through the secure Lime Survey-UV digital platform. Quantitative data will be analyzed using SPSS v29, following CONSORT guidelines. ANOVAs, χ² tests, and mixed-effects models will be used to analyze group-by-time interactions. Model fit indices for psychometric validation will be assessed using JASP. Qualitative data from focus groups will be analyzed thematically using NVivo or ATLAS.ti.

Collaborating Institutions:

University of Basque Country UPV/EUH

The principal investigators (Dr. Sandra Pérez and Dr. Monika Salgueiro) coordinate inter-university collaboration and oversight.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Be currently enrolled as a university student in a Spanish university.
* Have access to the internet via personal computer, smartphone, or tablet (only applicable for participation in the online format).
* Acknowledge that the program offered is a suicide prevention training intervention.
* Provide informed consent to participate.

Exclusion Criteria:

* Inability to understand Spanish (the program will be delivered exclusively in Spanish).
* Inability or unwillingness to commit to attending both training sessions (regardless of whether the participant ultimately continues in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in Willingness to Intervene Against Suicide (WISE) Score from Baseline to 2-Month Follow-Up | From baseline (T0) to T1 (2 weeks after T0), with a 2-3month follow-up at T2 (approximately 2.5 months after T0) and a follow-up at 9-12 months from T1 (T3)
  The Willingness to Intervene Against Suicide Enhanced Questionnaire (WISE) assesses four constructs from the Theory of Planned Behavior: (1) attitudes toward intervening in suicidal behavior, (2) subjective norms, (3) perceived behavioral control, and (4) intentions to intervene. The scale consists of multiple items rated on Likert-type scales. Higher scores indicate greater willingness and preparedness to act as a suicide prevention gatekeeper. The Spanish version of the WISE will be used, following a translation and back-translation process, and will be validated within this study.
Self-Reported Gatekeeper Behaviors Using ACT as Gatekeeper Scale from Baseline to 2-Month Follow-Up | From baseline (T0) to T1 (2 weeks after T0), with a 2-3month follow-up at T2 (approximately 2.5 months after T0) and a follow-up at 9-12 months from T1 (T3).
  The ACT as Gatekeeper scale evaluates the frequency of suicide prevention behaviors performed by participants over the previous three months. It includes five core actions: (1) asking someone about suicidal thoughts or emotional distress, (2) listening empathetically to a person in distress, (3) providing relevant information, (4) referring someone to an appropriate support resource, and (5) identifying suicide warning signs. Participants rate the frequency of each behavior. Higher scores indicate greater implementation of gatekeeper behaviors. The Spanish version of the instrument, translated and back-translated by the research team, will be validated as part of this study.

SECONDARY OUTCOMES:
Change in Suicide Literacy Score Using LOSS-SF from Baseline to 2-Month Follow-Up | From baseline (T0) to T1 (2 weeks after T0), with a 2-3month follow-up at T2 (approximately 2.5 months after T0) and a follow-up at 9-12 months from T1 (T3).
  The Literacy of Suicide Scale - Short Form (LOSS-SF) is a 12-item measure that assesses participants' knowledge and understanding of suicide. It evaluates four content areas: (1) causes and nature of suicide, (2) risk and protective factors, (3) warning signs, and (4) treatment and prevention. Each item is scored as correct or incorrect. Higher total scores reflect greater literacy about suicide. The study will use a Spanish version previously validated by Collado et al. (2023) and Pierantonelli et al. (2024).
Change in Stigma Toward Suicide Score Using SOSS-SF from Baseline to 2-Month Follow-Up | From baseline (T0) to T1 (2 weeks after T0), with a 2-3month follow-up at T2 (approximately 2.5 months after T0) and a follow-up at 9-12 months from T1 (T3)
  The Stigma of Suicide Scale - Short Form (SOSS-SF) includes 16 items measuring public attitudes toward individuals who die by suicide. Each item is a descriptor rated by the respondent and contributes to one of three subscales: (1) stigmatizing attitudes, (2) attribution of suicide to isolation or depression, and (3) normalization or glorification of suicide. Higher scores on the stigma subscale indicate more negative attitudes. A validated Spanish version will be used for this study.
Change in Depressive Symptoms Using PHQ-9 from Baseline to 2-Month Follow-Up | From baseline (T0) to T1 (2 weeks after T0), with a 2-3month follow-up at T2 (approximately 2.5 months after T0) and a follow-up at 9-12 months from T1 (T3)
  The PHQ-9 is a 9-item self-report questionnaire assessing depressive symptoms over the past two weeks, based on DSM-IV criteria. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. It has demonstrated good sensitivity (.87) and specificity (.88). The validated Spanish version (Diez-Quevedo et al., 2001) will be used.
Self-Reported Emotional Burden After Completing Gatekeeper Training | From baseline (T0) to T1 (2 weeks after T0), with a 2-3month follow-up at T2 (approximately 2.5 months after T0) and a follow-up at 9-12 months from T1 (T3)
  A single-item question assessing participants' emotional response to the training:
  "To what extent did participating in the program cause you emotional distress or stress?" Responses are rated on a 5-point Likert scale from 1 (Not at all) to 5 (Very much). This item provides insight into the psychological acceptability of the intervention.
Participant Satisfaction and Perceived Preparedness After Gatekeeper Training | Immediately after the training (T1): two weeks after T0.
  A short set of self-report questions assessing participants' satisfaction and perceived utility of the training. Items include:
  Global satisfaction with the training (1-10 scale). Willingness to recommend the program. Perceived preparedness to act as a gatekeeper (1-5 scale). One open-ended question on most useful aspects and suggestions for improvement.
Suicidal behavior (self and others) | From baseline (T0) to T1 (2 weeks after T0), with a 2-3month follow-up at T2 (approximately 2.5 months after T0) and a follow-up at 9-12 months from T1 (T3)
  Assessed through items examining personal history of suicidal ideation or attempts and exposure to suicidal behavior in close others (e.g., "Have you ever experienced suicidal thoughts?", "Has someone close to you attempted or died by suicide?"). These items were included to explore contextual and psychosocial correlates of preventive behavior, in line with the project protocol.
Intersession skill monitoring | After each training session.
  Captured through a 12-item self-report scale assessing progressive improvement in knowledge, attitudes, self-efficacy, behavioral intention, and detection-related actions after each training session (e.g., "After today's session, I feel more capable of recognizing warning signs", "I feel more confident in initiating a conversation with someone at risk").

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after deidentification
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available immediately following publication
Access Criteria: The data will be available to anyone who wishes to access them.

REFERENCES:
- [Result] Wolitzky-Taylor K, LeBeau RT, Perez M, Gong-Guy E, Fong T. Suicide prevention on college campuses: What works and what are the existing gaps? A systematic review and meta-analysis. J Am Coll Health. 2020 May-Jun;68(4):419-429. doi: 10.1080/07448481.2019.1577861. Epub 2019 Mar 25. PMID 30908123
- [Result] Litteken C, Sale E. Long-Term Effectiveness of the Question, Persuade, Refer (QPR) Suicide Prevention Gatekeeper Training Program: Lessons from Missouri. Community Ment Health J. 2018 Apr;54(3):282-292. doi: 10.1007/s10597-017-0158-z. Epub 2017 Aug 24. PMID 28840363
- [Result] Spafford SG, McWhirter Boisen MR, Tanner-Smith EE, Rodriguez G, Muruthi JR, Seeley JR. The Effects of Suicide Prevention Gatekeeper Training on Behavioral Intention and Intervention Behavior: A Systematic Review and Meta-Analysis. Prev Sci. 2024 Aug;25(6):978-988. doi: 10.1007/s11121-024-01710-w. Epub 2024 Jul 18. PMID 39023720
- [Result] Nozawa K, Ishii A, Asaoka H, Iwanaga M, Kumakura Y, Oyabu Y, Shinozaki T, Imamura K, Kawakami N, Miyamoto Y. Effectiveness of an Online Peer Gatekeeper Training Program for Postsecondary Students on Suicide Prevention in Japan: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Apr 26;11(4):e34832. doi: 10.2196/34832. PMID 35471412
- [Result] Pierantonelli M, Mira A, Zamora A, Desdentado L, Diego-Pedro R, Gonzalez-Hernandez E, Breton-Lopez J, Garcia-Palacios A, Banos RM. Levels and Predictors of Suicide Literacy and Suicide Stigma in Spanish-Speaking Individuals. Brain Behav. 2024 Nov;14(11):e70125. doi: 10.1002/brb3.70125. PMID 39501547
- [Result] Aldrich RS, Cerel J. The Willingness to Intervene Against Suicide Enhanced Questionnaire. Health Commun. 2024 Jul;39(8):1606-1615. doi: 10.1080/10410236.2023.2227435. Epub 2023 Jun 22. PMID 37349882
- [Result] Gould MS, Cross W, Pisani AR, Munfakh JL, Kleinman M. Impact of Applied Suicide Intervention Skills Training on the National Suicide Prevention Lifeline. Suicide Life Threat Behav. 2013 Dec;43(6):676-91. doi: 10.1111/sltb.12049. Epub 2013 Jul 25. Erratum In: Suicide Life Threat Behav. 2015 Apr;45(2):260. PMID 23889494